CLINICAL TRIAL: NCT01302054
Title: A 14 Week Randomized Parallel Group Placebo-Controlled Double-Blind Multicentre Study Of Fesoterodine 8 Mg In Overactive Bladder Patients With Sub-Optimal Response To Tolterodine 4 Mg Extended Release (ER).
Brief Title: A Clinical Study in Patients With Overactive Bladder With Leakage of Urine, to Find Out if the Medicine, Fesoterodine, Works in Those Patients Who Did Not Have Enough Response to the Medicine, Tolterodine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0221094
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Urinary Bladder, Overactive
Keywords: Bladder Overactive; Overactive urinary bladder; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fesoterodine (Experimental)
  Interventions: Drug: Fesoterodine 8 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fesoterodine 8 mg — Fesoterodine sustained release tablets once every morning at 4 mg dose for first week, followed by 11 weeks at 8 mg strength.
  Other Names: Toviaz
  Arms: Fesoterodine
Drug: Placebo — Matching placebo for fesoterodine 4 and 8 mg for a total of 12 weeks.
  Arms: Placebo

SUMMARY:
Patients with overactive bladder are often treated with tolterodine, a medication that helps relax the bladder, helping symptoms of urinary incontinence and urinary frequency. Sometimes patients do not have a satisfactory response, and may benefit from trying an alternative oral medicine. Fesoterodine is related to tolterodine by producing the same active substance that acts on the bladder, but potentially at higher and more effective levels. So, a patient who has a poor response to tolterodine may still obtain a good response to fesoterodine. This study will help find out if this is what happens.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder with symptoms for at least 6 months.
* Moderate to severe incontinence episode frequency and subsequent sub-optimal response to tolterodine
* Women of child-bearing potential must not intend to become pregnant, be pregnant or producing breast milk at the time of study entry, and must use contraception

Exclusion Criteria:

* Conditions or prior treatment that may also affect bladder function
* Clinically significant urinary tract infection (UTI)
* Ongoing treatment with overactive bladder medications (these can be stopped at the first visit to allow entry into the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (175):
- United States (109):
  - Radiant Research, Inc., Birmingham, Alabama
  - Alabama Internal Medicine, PC, Birmingham, Alabama
  - Brown and McCool Gynecology, Fairhope, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - Eclipse Clinical Research, Green Valley, Arizona
  - Radiant Research, Inc., Tucson, Arizona
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - American Institute of Research, Los Angeles, California
  - Moaz Khorsandi, DO, Los Angeles, California
  - Urology Group of Southern California, Los Angeles, California
  - Institute for Advanced Urology, Los Angeles, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Sierra Clinical Research, Roseville, California
  - Superior Research LLC, Sacramento, California
  - California Research Foundation, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Advanced Urology, PC, Parker, Colorado
  - Thameside Obstetrics/Gynecological Center, Groton, Connecticut
  - S.H.E. Medical Associates, Hartford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Manatee Medical Research Institute, LLC, Bradenton, Florida
  - Atlantic Institute of Clinical Research, Daytona Beach, Florida
  - SJS Clinical Research, Destin, Florida
  - Ocala Urology Specialists, Ocala, Florida
  - Renstar Medical Research, Inc., Ocala, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - Florida Urology Partners, Tampa, Florida
  - The Office of Georgis Patsias, MD, PA, Wellington, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Atlanta Medical Research Institute, LLC, Alpharetta, Georgia
  - Radiant Research, Inc., Atlanta, Georgia
  - In-Quest Medical Research, LLC, Duluth, Georgia
  - Prism Research Group, Rome, Georgia
  - Valley Health Care, Rome, Georgia
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - Radiant Research, Inc., Chicago, Illinois
  - Urology of Indiana, LLC, Noblesville, Indiana
  - Radiant Research, Inc., Overland Park, Kansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - New England Center for Clinical Research Fall River, LLC, Fall River, Massachusetts
  - New England Center for Clinical Research of Massachusetts, LLC, New Bedford, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - Medical Research Associates, Inc., Traverse City, Michigan
  - Radiant Research, Inc., Edina, Minnesota
  - Adult and Pediatric Urology, Sartell, Minnesota
  - CRC of Jackson, Jackson, Mississippi
  - Women's Specialty Center, Jackson, Mississippi
  - The Urology Group, Southaven, Mississippi
  - Radiant Research, Inc., St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Francis Jimenez, MD, Las Vegas, Nevada
  - Impact Clinical Trials, Las Vegas, Nevada
  - Richard M. Groom, MD, Las Vegas, Nevada
  - Northeast Urogynecology, Albany, New York
  - The Urologic Institute of Northeastern New York - Community Care Physicians, PC, Albany, New York
  - University Urology Associates, New York, New York
  - Associated Medical Professionals of New York, PLLC, Oneida, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Urology Specialists of the Carolinas, Charlotte, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Salibury Urological Clinic, Salisbury, North Carolina
  - Carolina Urological Associates, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Radiant Research, Inc., Akron, Ohio
  - Radiant Research, Inc., Cincinnati, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Pacific Women's Center, LLC, Eugene, Oregon
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - OB/GYN Associates of Erie, Erie, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Gilbert Teixeira, DO, East Providence, Rhode Island
  - Pharma Resource, East Providence, Rhode Island
  - Memorial Hospital of Rhode Island - Clinical Studies Center, Pawtucket, Rhode Island
  - Radiant Research, Inc., Anderson, South Carolina
  - Columbia Women's Healthcare, LLC, Columbia, South Carolina
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - OB-GYN Centre of Excellence, Chattanooga, Tennessee
  - Advanced Therapeutics, Inc., Johnson City, Tennessee
  - Johnson City Internal Medicine, Johnson City, Tennessee
  - Adult Care of Austin, Austin, Texas
  - Senior Adults Specialty Research, Austin, Texas
  - DiscoveResearch, Inc., Beaumont, Texas
  - Beaumont Internal Medicine & Geriatric Associates, Beaumont, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - DiscoveResearch, Incorporated, Bryan, Texas
  - Radiant Research, Inc., Dallas, Texas
  - Advances In Health, Inc., Houston, Texas
  - Centex Research, Inc. - Pineloch Medical Clinic, Houston, Texas
  - The Office of Dr. Steven Maislos, MD, Houston, Texas
  - Village Health Partners, Plano, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Radiant Research, Inc., Murray, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Integra Trials, LLC, Arlington, Virginia
  - Washington Urology, Arlington, Virginia
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington
  - Urology Northwest, PA, Mountlake Terrace, Washington
  - North Spokane Women's Clinic, Spokane, Washington
- Bulgaria (5):
  - MBAL Trimontsium OOD, Plovdiv
  - MBAL Ruse AD, Urologichno otdelenie,, Rousse
  - UMBAL Aleksandrovska EAD, Sofia
  - MBALSM N.I.Pirogov EAD, Sofia
  - MBAL Doverie AD, Otdelenie po urologia, Sofia
- Canada (10):
  - The Prostate Cancer Centre, Calgary, Alberta
  - Lois Hole Hospital for Women, Royal Alexandra Hospital, Edmonton, Alberta
  - Maritime Research Center, Bathurst, New Brunswick
  - The Male/Female Health and Research Centre, Royal Court Medical Centre, Barrie, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Centre for Applied Urological Research, Queen's University, Kingston General Hospital, Kingston, Ontario
  - URLX Corporation, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Diex Research Montreal Inc., Montreal, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Czechia (4):
  - Prvni privatni chirurgicke centrum spol. s .r.o. - SANUS, Hradec Králové
  - Nemocnice Jindrichuv Hradec, Jindřichův Hradec
  - Oblastni nemocnice Kolin, a.s., Kolin III
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- Ain Shams University Hospital, Cairo, Egypt
- Suomen Terveystalo Turku, Turku, Finland
- Germany (11):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Klinische Forschung Berlin, Berlin
  - Praxis fuer Urologie, Berlin
  - Duisburger Fachaerztegemeinschaft, Duisburg
  - ZKS Suedbrandenburg GmbH, Elsterwerda
  - Facharzt für Frauenheilkunde und Geburtshilfe, Frankfurt am Main
  - Urologische Praxis, Hagenow
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Arztpraxis Dr. von Keitz, Marburg
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Mittweida
  - Frauenarzt Praxis, München
- Hungary (4):
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar Urologiai Klinika, Budapest
  - Soproni Erzsebet Oktato Korhaz, Urologiai Osztaly, Sopron
  - Donatella 99 Bt., Szentes
  - MAV Korhaz es Rendelointezet, Urologia, Szolnok
- Mexico (2):
  - Phylasis Clinicas Research S de RL de CV, Cuautitlán Izcalli, State of Mexico
  - Unidad de Diagnostico Integral, Colima
- Poland (3):
  - NZOZ VIP - MED, Poradnia Urologiczna, Gdynia
  - SP ZOZ Wojewodzki Szpital Specjalistyczny im. J. Koraczaka, Słupsk
  - Specjalistyczny Gabinet Lekarski, Warsaw
- Russia (7):
  - Kemerovо Regional Perinatal Center, Kemerovo
  - Moscow State Healthcare Institution City Clinical Hospital #12, Moscow
  - Saint-Petersburg State Budgetary Healthcare Institution City Hospital #26, Saint Petersburg
  - Saint-Petersburg State Medical University I.P.Pavlov, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution City Hospital # 15, Saint Petersburg
  - St. Petersburg State Healthcare Institution, Saint Petersburg
  - Siberian State Medical University, Tomsk
- Parklands Hospital, Durban, KwaZulu-Natal, South Africa
- South Korea (3):
  - Department of Urology, Pusan National University Hospital, Pusan
  - Department of Urology, Konkuk University Medical Center, Seoul
  - Department of Urology, Ajou University Hospital, Suwon
- Sweden (6):
  - Kvinnohalsan Soder, Bandhagen
  - Specialistmottagningen i urologi, Gothenburg
  - Partus Kvinnohalsa, Gothenburg
  - Me3plus Clinical Trials, Gothenburg
  - Tudorkliniken, Specialistmottagningen i Urologi, Halmstad
  - Vrinnevisjukhuset, Norrköping
- Ukraine (8):
  - Regional Clinical Hospital, Department of Urology of Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Regional Clinical Center of Urology and Nephrology, Kharkiv
  - Institute of Urology of AMS of Ukraine, Kyiv
  - Lugansk City Multi-Discipline Hospital #2, department of Urology, Luhansk
  - 5Th City Clinical Hospital, Urology Department, Lviv
  - LTD Out-patient clinic of General practice and Family medicine, Odesa
  - Poltava Regional Clinical Hospital, Department of Urology, Poltava
  - Municipal Institution of Ternopil Regional Council, Ternopil University Hospital, Ternopil

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Wagg AS, Herschorn S, Carlsson M, Fernet M, Oelke M. A plain language summary of the likelihood of symptom relief for patients taking fesoterodine for overactive bladder. J Comp Eff Res. 2022 Sep;11(13):919-925. doi: 10.2217/cer-2022-0041. Epub 2022 Jul 26. PMID 35881009
- [Derived] Kaplan SA, Cardozo L, Herschorn S, Grenabo L, Carlsson M, Arumi D, Crook TJ, Whelan L, Scholfield D, Ntanios F; Assessment of Fesoterodine after Tolterodine ER (AFTER) Study Group. Efficacy and safety of fesoterodine 8 mg in subjects with overactive bladder after a suboptimal response to tolterodine ER. Int J Clin Pract. 2014 Sep;68(9):1065-73. doi: 10.1111/ijcp.12464. Epub 2014 Jun 4. PMID 24898471
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221094

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolterodine: Tolterodine 4 milligram (mg) extended release capsule orally once daily for 2 weeks during open-label run-in phase. Participants who were non-responders in the open-label run-in phase (defined as participants who had less than or equal to [<=] 50 percent change in urgency urinary incontinence [UUI] episodes), were randomized to either fesoterodine or placebo group, in double-blind treatment phase.
- Fesoterodine: Fesoterodine 4 mg sustained release tablet orally once daily for 1 week followed by fesoterodine 8 mg sustained release tablet orally once daily up to Week 12 during double-blind treatment phase.
- Placebo: Matching placebo tablet orally once daily for 12 weeks during double-blind treatment phase.
Period: Tolterodine Open-Label Run-In Phase
Arm/Group | Tolterodine | Fesoterodine | Placebo
Started | 990 | 0 | 0
Completed | 611 | 0 | 0
Not Completed | 379 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Lost to Follow-up | 17 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 0
Not completed — Adverse Event | 13 | 0 | 0
Not completed — Did Not Meet Entrance Criteria | 314 | 0 | 0
Not completed — Other | 7 | 0 | 0
Period: Between Open-Label and Double Blind
Arm/Group | Tolterodine | Fesoterodine | Placebo
Started | 611 | 0 | 0
Completed | 609 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Did Not Enter Double-Blind Phase | 2 | 0 | 0
Period: Double-Blind Treatment Phase
Arm/Group | Tolterodine | Fesoterodine | Placebo
Started | 0 | 308 | 301
Completed | 0 | 281 | 255
Not Completed | 0 | 27 | 46
Not completed — Lack of Efficacy | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 14
Not completed — Protocol Violation | 0 | 3 | 6
Not completed — Adverse Event | 0 | 10 | 10
Not completed — Did Not Meet Entrance Criteria | 0 | 0 | 2
Not completed — Other | 0 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Tolterodine 4 milligram (mg) extended release capsule orally once daily for 2 weeks during open-label run-in phase. Participants who were non-responders in the open-label run-in phase (defined as participants who had <= 50 percent change in UUI episodes), were randomized to either fesoterodine or placebo group, in double-blind treatment phase.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 990
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 810
  Male | 180

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours
Description: UUI episodes were defined as those with the urinary sensation scale (USS) rating of 5 in the diary. USS range from 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Week 12
Population: Full analysis set:all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Last Observation Carried Forward(LOCF) was used. N(number of participants analyzed):participants with baseline UUI episodes >0 per 24 hours and non-missing change from baseline at Week 12(LOCF).
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Groups:
- Fesoterodine: Double-Blind Baseline: Participants who were randomized to receive fesoterodine 4 mg sustained release tablet orally once daily for 1 week followed by fesoterodine 8 mg sustained release tablet orally once daily up to Week 12 during double-blind treatment phase.
- Fesoterodine: Double-Blind Week 12: Participants who received fesoterodine 4 mg sustained release tablet orally once daily for 1 week followed by fesoterodine 8 mg sustained release tablet orally once daily up to Week 12 during double-blind treatment phase.
Arm/Group | Fesoterodine: Double-Blind Baseline | Fesoterodine: Double-Blind Week 12
Number analyzed (Participants) | 292 | 292
episodes per 24 hours | 3.93 (2.53) | 1.60 (2.56)
Statistical Analysis 1: Comparison: Fesoterodine: Double-Blind Baseline vs Fesoterodine: Double-Blind Week 12; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — Statistical testing: one-sided, at alpha = 0.025; Least Squares Mean Difference = -2.37, 95% CI 2-sided [-2.63 to -2.02], Standard Error of Mean 0.17

2. Primary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Full Analysis set (FAS): all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Missing data were imputed by LOCF. N (number of participants analyzed): participants with baseline UUI episodes >0 per 24 hours and non-missing change from baseline at Week 12 (LOCF).
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 292 | 279
episodes per 24 hours
  Baseline | 3.93 (2.53) | 3.83 (2.52)
  Change at Week 12 | -2.32 (2.67) | -1.76 (2.46)
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Multiple hypothesis testing was carried out in a hierarchical sequentially rejective manner. Statistical testing between fesoterodine and placebo (Analysis of covariance [ANCOVA]) was carried out only if the change from baseline at Week 12 in UUI episodes for fesoterodine group was found statistically significant (paired t-test); Test type: Superiority or Other; p = 0.0079, ANCOVA — Change at Week 12: ANCOVA model with terms for treatment and country with centered baseline value as a covariate was used. Statistical testing: one-sided, at alpha = 0.025; Least Squares Mean Difference = -0.50, 95% CI 2-sided [-0.87 to -0.13], Standard Error of Mean 0.19

3. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 12
Description: Micturitions include episodes of voluntary micturition and episodes of Urgency Urinary Incontinence (UUI). UUI episodes were defined as those micturitions with USS rating of 5 in the diary in participants with UUI at baseline. USS rating 5: Unable to hold; leak urine.
Time Frame: Baseline, Week 12
Population: FAS: all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Missing data were imputed by LOCF. Here 'N' (number of participants analyzed): participants with baseline micturitions >0 per 24 hours and non-missing change from baseline at Week 12 (LOCF).
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 292 | 279
micturitions per 24 hours
  Baseline | 12.44 (3.57) | 12.48 (3.75)
  Change at Week 12 | -1.94 (3.15) | -1.57 (3.13)
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Change at Week 12: ANCOVA model with terms for treatment and country with centered baseline value as a covariate was used; Test type: Superiority or Other; p = 0.0931, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; Least Squares Mean Difference = -0.40, 95% CI 2-sided [-0.86 to 0.07], Standard Error of Mean 0.24

4. Secondary Outcome: Change From Baseline in Mean Number of Micturition-Related Urgency Episodes Per 24 Hours at Week 12
Description: The mean number of micturition-related urgency episodes per 24 hours was calculated as the total number of micturitions with USS rating of greater than or equal to 3 divided by the total number of days that diary data was collected at that visit. USS range from 1 to 5: 1. No feeling of urgency, 2. Mild feeling of urgency, 3. Moderate feeling of urgency, 4. Severe feeling of urgency, 5. Unable to hold; leak urine.
Time Frame: Baseline, Week 12
Population: FAS: all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Missing data were imputed by LOCF. Here 'N' (number of participants analyzed): participants with baseline urgency episodes >0 per 24 hours and non-missing change from baseline at Week 12 (LOCF).
Measure: Mean (Standard Deviation); unit: episodes per 24 hours
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 292 | 279
episodes per 24 hours
  Baseline | 11.38 (3.98) | 11.26 (4.01)
  Change at Week 12 | -3.33 (4.47) | -2.52 (4.45)
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0438, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; Least Squares Mean Difference = -0.70, 95% CI 2-sided [-1.37 to -0.02], Standard Error of Mean 0.34

5. Secondary Outcome: Number of Participants With Change From Baseline in Patient Perception of Bladder Condition (PPBC) at Week 12
Description: PPBC: single-item, self-administered validated questionnaire. Participant answered: "Which of the following statements describes your bladder condition best at the moment?" on a 6-point scale, 1=no problems at all; 2=some very minor problems; 3=some minor problems; 4=some moderate problems; 5=severe problems; 6=many severe problems. Change=observation minus baseline. Results categorized as Deterioration (Positive change from baseline); No Change (scores change=0); Minor Improvement (negative score change in magnitude of 1); Major Improvement (negative score change in magnitude of >=2).
Time Frame: Baseline, Week 12
Population: FAS: all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Here, 'N' (number of participants analyzed): participants with non-missing change from baseline value at Week 12.
Measure: Number; unit: participants
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 291 | 267
participants
  Baseline: No Problems at all | 0 | 0
  Baseline: Some Very Minor Problems | 4 | 6
  Baseline: Some Minor Problems | 15 | 9
  Baseline: Some Moderate Problems | 60 | 75
  Baseline: Severe Problems | 147 | 141
  Baseline: Many Severe Problems | 65 | 36
  Change at Week 12: Deterioration | 17 | 32
  Change at Week 12: No Change | 80 | 95
  Change at Week 12: Minor Improvement | 84 | 83
  Change at Week 12: Major Improvement | 110 | 57
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Change at Week 12: the p-value was obtained from a Cochran-Mantel-Haenszel (CMH) test with modified ridit scoring controlling for country

6. Secondary Outcome: Number of Participants With Change From Baseline in Urgency Perception Scale (UPS) at Week 12
Description: UPS: single-item, self-administered validated questionnaire. Participant answered: "Which of the following would typically describe your experience when you have a desire to urinate?" on a 3-point scale, 1=usually not able to hold urine; 2=usually able to hold urine (without leaking) until I reach a toilet if I go to the toilet immediately; 3= usually able to finish what I am doing before going to the toilet (without leaking). Change = observation minus baseline. Results categorized as Deterioration (Negative change); no change (Score change=0); improvement (Positive change).
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 291 | 267
participants
  Baseline: Not able to hold urine | 126 | 99
  Baseline:Able to hold urine until I reach a toilet | 158 | 157
  Baseline:Able to finish what I am doing | 7 | 11
  Change at Week 12: Deterioration | 17 | 31
  Change at Week 12: No Change | 167 | 158
  Change at Week 12: Improvement | 107 | 78
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Test type: Superiority or Other; p = 0.0095, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score at Week 12
Description: OAB-q: a self-administered, 33-item, questionnaire that assesses how much the participant has been bothered by selected bladder symptoms. Each item rated by participant on Likert scale 1 (not at all) to 6 (a very great deal). Symptom bother score derived as sum of scores for questions 1-8; lowest possible raw score: 8; highest possible score: 48. Data analyzed based on transformation of the score to a 0 to 100 scale [(Actual total raw score - lowest possible value of raw score)/range]*100. Higher scores values indicative of greater symptom bother. Change=observation minus baseline.
Time Frame: Baseline, Week 12
Population: FAS: all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Here 'N' (number of participants analyzed): participants with non-missing change from baseline value at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 286 | 267
units on a scale
  Baseline | 66.67 (20.28) | 64.74 (19.69)
  Change at Week 12 | -24.61 (25.57) | -15.99 (24.53)
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; Least Squares Mean Difference = -7.34, 95% CI 2-sided [-11.10 to -3.58], Standard Error of Mean 1.91

8. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQL) Domains and Total HRQL Score of Overactive Bladder Questionnaire (OAB-q) at Week 12
Description: OAB-q: self-administered, 33-item, questionnaire, assesses how much participant has been bothered by selected bladder symptoms. Each item rated on Likert scale 1 (not at all) to 6 (a very great deal). Questions 9 to 33 constitute HRQL, includes domains: concern, coping, sleep, and social function. HRQL domain and total raw score derived as sum of scores. Transformed score range 0 to 100 (Total HRQL or domain) = [(Highest possible raw score-Actual total raw score)/Raw score range]*100. Higher transformed scores indicative of better HRQL.
Time Frame: Baseline, Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 286 | 267
units on a scale
  Concern Subscale: Baseline | 43.63 (26.00) | 44.25 (25.58)
  Concern Subscale: Change at Week 12 | 23.11 (27.77) | 13.83 (25.03)
  Coping Subscale: Baseline | 38.74 (26.24) | 41.15 (26.04)
  Coping Subscale: Change at Week 12 | 23.70 (26.69) | 15.07 (24.20)
  Sleep Subscale: Baseline | 41.38 (25.66) | 40.69 (26.28)
  Sleep Subscale: Change at Week 12 | 20.85 (27.42) | 14.79 (25.74)
  Social Interaction Subscale: Baseline | 65.03 (28.34) | 68.40 (26.29)
  Social Interaction Subscale: Change at Week 12 | 14.47 (24.26) | 8.85 (21.12)
  Total HRQL Score: Baseline | 45.90 (23.72) | 47.38 (22.70)
  Total HRQL Score: Change at Week 12 | 21.12 (24.62) | 13.42 (21.92)
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Concern Subscale - Change at Week 12: ANCOVA model with terms for treatment and country with centered baseline value as a covariate was used; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; Least Squares (LS) Mean Difference = 9.01, 95% CI 2-sided [5.12 to 12.91], Standard Error of Mean 1.98
Statistical Analysis 2: Comparison: Fesoterodine vs Placebo; Coping Subscale - Change at Week 12: ANCOVA model with terms for treatment and country with centered baseline value as a covariate was used; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; LS Mean Difference = 7.75, 95% CI 2-sided [3.87 to 11.62], Standard Error of Mean 1.97
Statistical Analysis 3: Comparison: Fesoterodine vs Placebo; Sleep Subscale - Change at Week 12: ANCOVA model with terms for treatment and country with centered baseline value as a covariate was used; Test type: Superiority or Other; p = 0.0012, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; LS Mean Difference = 6.52, 95% CI 2-sided [2.60 to 10.45], Standard Error of Mean 2.00
Statistical Analysis 4: Comparison: Fesoterodine vs Placebo; Social Interaction Subscale - Change at Week 12: ANCOVA model with terms for treatment and country with centered baseline value as a covariate was used; Test type: Superiority or Other; p = 0.0123, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; LS Mean Difference = 4.13, 95% CI 2-sided [0.90 to 7.36], Standard Error of Mean 1.64
Statistical Analysis 5: Comparison: Fesoterodine vs Placebo; Total HRQL - Change at Week 12: ANCOVA model with terms for treatment and country with centered baseline value as a covariate was used; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing: one-sided, at alpha = 0.025; LS Mean Difference = 7.10, 95% CI 2-sided [3.63 to 10.57], Standard Error of Mean 1.77

9. Secondary Outcome: Percentage of Participants With More Than (>) 50 Percent (%) Reduction in UUI Episodes at Week 12 as Compared to Week -2
Description: as for outcome 1
Time Frame: Week -2, Week 12
Population: FAS: all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Missing data were imputed by LOCF. N (number of participants analyzed): participants with Week -2 UUI episodes >0 per 24 hours and non-missing change from baseline at Week 12 (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 279 | 275
percentage of participants | 72.8 | 59.6
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Test type: Superiority or Other; p = 0.0023, Cochran-Mantel-Haenszel — The p-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test and stratified by country

10. Secondary Outcome: Percentage of Participants With More Than (>) 50 Percent (%) Reduction in UUI Episodes at Week 12 as Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: FAS: all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Missing data were imputed by LOCF. N (number of participants analyzed): participants with baseline UUI episodes >0 per 24 hours and non-missing change from baseline at Week 12 (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 292 | 279
percentage of participants | 69.9 | 57.0
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Test type: Superiority or Other; p = 0.0027, Cochran-Mantel-Haenszel — The p-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test and stratified by country

11. Secondary Outcome: Percentage of Participants With No UUI Episodes (Diary Dry Rate)
Description: as for outcome 1
Time Frame: Week 4, Week 12
Population: FAS: all randomized participants who received at least 1 dose of double-blind study treatment, had baseline/post-baseline efficacy assessment. Missing data were imputed by LOCF. N (number of participants analyzed): participants with baseline UUI episodes >0 per 24 hours and non-missing change from baseline at Week 4 and 12 (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Fesoterodine | Placebo
Number analyzed (Participants) | 292 | 279
percentage of participants
  Week 4 | 25.4 | 17.7
  Week 12 | 39.0 | 32.3
Statistical Analysis 1: Comparison: Fesoterodine vs Placebo; Test type: Superiority or Other; p = 0.0427, Cochran-Mantel-Haenszel — Treatment difference at Week 4: p-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test and stratified by country
Statistical Analysis 2: Comparison: Fesoterodine vs Placebo; Test type: Superiority or Other; p = 0.1461, Cochran-Mantel-Haenszel — Treatment difference at Week 12: p-value was obtained from a Cochran-Mantel-Haenszel (CMH) general association test and stratified by country

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tolterodine | Fesoterodine | Placebo
Serious Adverse Events (participants affected / at risk) | 3/990 | 5/308 | 7/301
Other Adverse Events (participants affected / at risk) | 90/990 | 76/308 | 48/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolterodine (N=990) | Fesoterodine (N=308) | Placebo (N=301)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolterodine (N=990) | Fesoterodine (N=308) | Placebo (N=301)
Vision blurred (Eye disorders) | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 11 | 12 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 4
Dry mouth (Gastrointestinal disorders) | 61 | 51 | 12
Dyspepsia (Gastrointestinal disorders) | 2 | 6 | 0
Nausea (Gastrointestinal disorders) | 7 | 1 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 4
Influenza (Infections and infestations) | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 6 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 3
Urinary tract infection (Infections and infestations) | 3 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 4
Headache (Nervous system disorders) | 4 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.